CLINICAL TRIAL: NCT04176822
Title: The Effects of Designing an Educational Animated Movie About Preoperative Preparation on Fear and Post-Operative Pain in Children:A Randomized Controlled Trial
Brief Title: Designing Animated Movie for Preoperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Şeyda BİNAY YAZ, Principal Investigator, Assistant Professor, PhD, Ege University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: SYaz; Ege (Other: Ege University)
Record Dates: First submitted 2019-11-01; First posted 2019-11-25 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain; Fear; Surgery; Pain; Nursing Caries; Nurse's Role; Clinical Anxiety; Patient; Pediatric
Keywords: pediatric surgery; preoperative preparation; animation; fear; pain; nursing
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: There are 3 independent working groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Educational Animated Movie Group (Experimental): All of the children's and parents' written and verbal informed consent were obtained before the study. Parents who did not want to participate in the study were assured that this would not have any adverse effect on their child's treatment. In the morning of surgery, the researcher administered the "Child and Family Identification Data Form" to the parents of children who had the following parameters. Later, both the child and the parents were asked to complete the "Children's Fear Scale". Children included in the study groups with randomization watched an educational animated movie through VR Goggles. The educational animated movie lasted around 3-4 minutes each. After watching the movie, children and parents were asked to complete the Children's Fear Scale again. Children, parents, and nurses were asked to grade the pain of the child with Wong-Baker FACES Pain Rating Scale when the children returned to their room and after 1 hour in the postoperative period.
  Interventions: Other: Educational animated movie group
- Documentary Movie Group (Experimental): All of the children's and parents' written and verbal informed consent were obtained before the study. Parents who did not want to participate in the study were assured that this would not have any adverse effect on their child's treatment. In the morning of surgery, the researcher administered the "Child and Family Identification Data Form" to the parents of children who had the following parameters. Later, both the child and the parents were asked to complete the "Children's Fear Scale". Children included in the study groups with randomization watched a documentary movie through VR Goggles. The documentary movie lasted around 3-4 minutes each. After watching the movie, children and parents were asked to complete the Children's Fear Scale again. Children, parents, and nurses were asked to grade the pain of the child with Wong-Baker FACES Pain Rating Scale when the children returned to their room and after 1 hour in the postoperative period.
  Interventions: Other: Documentary movie group
- Control Group (No Intervention): No intervention was made, pain and fear levels were measured using scales only.

INTERVENTIONS:
Other: Educational animated movie group — Watching educational animation movie which were designed by the researcher before operation for fear and pain.
  Arms: Educational Animated Movie Group
Other: Documentary movie group — Watching documentary movie about trees before operation for fear and pain.
  Arms: Documentary Movie Group

SUMMARY:
Background: Using visual materials is effective in education to decrease children's pre-operative fear and post-operative pain. Children, especially those aged between 6 and 12 years, are interested in technology. This study aims to investigate the effects of watching an educational animated movie in the pre-operative period on fear and postoperative pain in children who are having surgery.

Methods: The study was a prospective randomized controlled trial. This study was conducted between 6- to 12-year-old children in the Pediatric Surgery Clinic of Ege University Medical Faculty Hospital. The current study includes data from 132 children who were chosen doing block randomization. The "Child and Family Identification Data Form", "Children's Fear Scale" and "Wong-Baker FACES Pain Rating Scale" was used in data collection. The patients were divided randomly into three groups as the "Educational Animated Movie Group" (EAMG), "Documentary Movie Group" (DMG) and "Control Group" (CG). The Educational Animated Movie and Documentary Movie were screened using Virtual Reality (VR). Data were collected by the researcher in the pre-operative period. The pre-operative fear of the child was evaluated by the child and the parent, and the post-operative pain of the child was evaluated by the child, parent, and nurse using scales about fear and pain.

ELIGIBILITY:
Inclusion Criteria:

* First surgery
* Daily surgery and uncomplicated surgery
* Agree to participate in the study
* Speaking Turkish

Exclusion Criteria:

* Refusal to participate in the study
* A genetic/congenital disease
* A chronic disease
* Second or more surgery
* Not speaking Turkish

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Change of Children's Preoperative Fear | 15 minutes (2 measurements are made-before and after intervention)
  "Children's Fear Scale" (CFS) was developed and adapted by McMurtry et al. (2011).
  This scale includes 5 different facial expressions. This scale, graded between 0 and 4, ("0" is none fear, "4" is maximum fear) is a reliable and valid measurement tool for assessing fear.
  It includes measuring and evaluating preoperative fears of children.
Change of Children's Postopeartive Pain | 15 minutes (2 measurements are made-immediately after surgery and 1 hour after surgery) = total 90 minutes
  "Wong-Baker FACES Pain Rating Scale" This scale includes six different facial expressions and is scored between 0 and 10 ("0" is none pain, "10" is maximum pain). It is a reliable and valid measurement tool for acute pain assessment, and it does not require words or numeric value.
  It includes measuring and evaluating postoperative pains of children.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study will be prepared for publication